CLINICAL TRIAL: NCT06165640
Title: Dietary Sodium Intake in Children on Chronic Dialysis: A Collaborative Study With the European Pediatric Dialysis Working Group
Brief Title: Dietary Sodium Intake in Children on Chronic Dialysis
Acronym: PeDialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8171
Record Dates: First submitted 2022-12-13; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2022-12

CONDITIONS: Chronic Dialysis in Children
Keywords: Chronic Dialysis in Children; Cardiovascular Diseases; Renal Diseases; Left Ventricular Hypertrophy; Hemodialysis Complication
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease is common in patients with end-stage renal disease that began in childhood, and volume overload plays a key role in the development of hypertension, left ventricular hypertrophy (LVH) and alterations. cardiovascular disease in this population. Thus, inter-dialytic weight gain is correlated with blood pressure and left ventricular mass index in children on hemodialysis (HD). Significant inter-dialytic weight gain in dialysis patients is largely due to thirst secondary to salt ingestions: attempts at water restriction without concomitant sodium restriction will probably be in vain. Additionally, sodium overload negatively affects blood pressure and cardiovascular status through various mechanisms unrelated to volume expansion.

Soda extraction by dialysis is often difficult, and sodium control is largely dependent on restricting dietary sodium intake. Some studies in adults have shown that a low sodium diet reduced inter-dialytic weight gain, reduced intra-dialytic complications, improved blood pressure values, and lowered index. left ventricular mass and mortality in dialysis patients.

For children with chronic kidney disease, data from the American Chronic Kidney Disease (CKiD) study show that the median sodium intake in children without dialysis with chronic kidney disease exceeds the maximum recommended intakes for all patients. age groups.

No study to date has investigated the average dietary sodium intake of children on dialysis. And, more importantly, the relationship between dietary sodium intake and cardiovascular morbidity has never been studied in children on dialysis.

ELIGIBILITY:
Inclusion Criteria :

* Minor patient (≥ 3 months and <18 years)
* Under the care of the University Hospitals of Strasbourg
* Having benefited from chronic dialysis (> 3 months)
* Having undergone hemodialysis (HD) or hemodiafiltration (HDF), 3 sessions / week, or automated peritoneal dialysis (PD)
* Subject (and / or his parental authority) not having expressed, after being informed, his opposition to the reuse of his data for the purposes of this research.

Non-Inclusion Criteria :

* Patient or one of the parents who expressed their opposition to participating in the study
* Intensive hemodialysis (HD at home, HD at night, ≥ 4 sessions / week)
* Intercurrent illness or clinical instability (left to the judgment of the physician)
* Non-nephrological diseases causing loss of salt (eg cystic fibrosis, etc.)
* Any physical or psychosocial situation that prevented the 24-hour ambulatory BP measurement from being taken, or poor compliance with the dietetic collection, etc.).

Ages: 3 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Minor patient (≥ 3 months and <18 years) having benefited from chronic dialysis (> 3 months) and having undergone hemodialysis (HD) or hemodiafiltration (HDF), 3 sessions / week, or automated peritoneal dialysis (PD) at the University Hospitals of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the average dietary intake of sodium (Na+) in a population of children on chronic dialysis. | Files analysed retrospectively from January 1, 2019 to February 28, 2021 will be examined
  The average dietary intake of sodium (Na+) is calculated according to the formula: sodium salt content (g) = Sodium (g) × 2.54

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France